CLINICAL TRIAL: NCT02472574
Title: Phase 2 Study of Rt-PA Dose-effect Relationship on ICH Evacuation
Brief Title: Dose-effect Relationship of Rt-PA on ICH Evacuation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Suiqiang Zhu, director of the neurology, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150403
Record Dates: First submitted 2015-05-17; First posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Hypertensive Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; minimally invasive surgery; recombinant tissue plasminogen activator; Dose-effect Relationship
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive; Cerebral Hemorrhage | interventions — Suction; Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.3 mg (Experimental): Subjects randomized to the 0.3 mg arm will undergo minimally invasive surgery with YL-1 type of intracranial hematoma puncture needle, followed by up to 4 doses of 0.3 mg of rt-PA (Activase/Alteplase/CathFlo) for intracerebral hemorrhage clot resolution.
  Interventions: Device: YL-1 type of intracranial hematoma puncture needle; Drug: rt-PA
- 0.5 mg (Experimental): Subjects randomized to the 0.5 mg arm will undergo minimally invasive surgery with YL-1 type of intracranial hematoma puncture needle,followed by up to 4 doses of 0.5 mg of rt-PA (Activase/Alteplase/CathFlo) for intracerebral hemorrhage clot resolution.
  Interventions: Device: YL-1 type of intracranial hematoma puncture needle; Drug: rt-PA
- 1.0 mg (Experimental): Subjects randomized to the 1.0 mg arm will undergo minimally invasive surgery with YL-1 type of intracranial hematoma puncture needle,followed by up to 4 doses of 1.0 mg of rt-PA (Activase/Alteplase/CathFlo) for intracerebral hemorrhage clot resolution.
  Interventions: Device: YL-1 type of intracranial hematoma puncture needle; Drug: rt-PA

INTERVENTIONS:
Device: YL-1 type of intracranial hematoma puncture needle — YL-1 type of intracranial hematoma puncture needle(Pat. NO.is ZL：93244252•8) was originated by Beijing WanTeFu Medical Apparatus Co.Ltd in 1997. With integration of needle and bur drill it is designed as hard tunnel.By the technique of skull self-holding, the puncture needle can being fixed in the target of haematoma for several days.This technique is convenient, simple and safe. To position haematoma's location, drills 3 millimeter holes in the localization point of puncture, then insert the drainage tube to inhale hematoma, gives the filament resolver interrupted for liquefication drainage afterward.
  Other Names: aspiration drainage
Drug: rt-PA — Up to 4 doses of 0.3~1.0 mg of rt-PA will be administered through the catheter that was placed directly into the intracerebral hemorrhage using minimally invasive surgery.
  Other Names: recombinant tissue plasminogen activator

SUMMARY:
The purpose of this trial is to determine the optimal dose of rt-PA in the treatment of intracerebral hemorrhage (ICH) using a combination of minimally invasive surgery and clot lysis with rt-PA。

DETAILED DESCRIPTION:
The minimally invasive surgery (MIS) plus recombinant tissue plasminogen activator (rt-PA) is one of the best choices in the treatment of a large-scale deep supratentorial intracerebral hematoma. It uses hardware access technology, in a relatively short time to enter the hematoma center with favourable accuracy and safety.

The dose of rt-PA range from 0.3 mg to 4.0 mg in different research。We propose to determine the optimal dose of rt-PA with three dose control groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80.
* GCS < 14 or a NIHSS > or equal to 6.
* Spontaneous supratentorial ICH ≥ 20 mL diagnosed using radiographic imaging (CT, CTA, etc.)
* Symptoms less than 24 hours prior to diagnostic CT(dCT) scan (an unknown time of symptom onset is exclusionary).
* Six-hour clot size equal to the most previous clot size (within 5 mL) as determined by additional CT scans at least 6 hours apart using the ABC/2 method.
* Intention to initiate surgery between 12 and 72 hours after after diagnostic CT. First dose can be given within 76 hours after dCT (delays for post surgical stabilization of catheter bleeding).
* SBP < 180 mmHg sustained for 6 hours recorded closest to time of randomization.
* Historical Rankin score of 0 or 1.
* Negative pregnancy test.

Exclusion Criteria:

* Infratentorial hemorrhage (any involvement of the midbrain or lower brainstem as demonstrated by radiograph or complete third nerve palsy).
* Irreversible impaired brain stem function (bilateral fixed, dilated pupils and extensor motor posturing), GCS ≤ 4.
* Intraventricular hemorrhage requiring treatment with extraventricular drainage (obstruction of third and fourth ventricles).
* Ruptured aneurysm, arteriovenous malformation (AVM), vascular anomaly, Moyamoya disease diagnosed with radiographic imaging.
* Any irreversible coagulopathy or known clotting disorder. or having the experience of the use of anticoagulant drug.
* Platelet count < 100,000, INR > 1.7, or an elevated prothrombin time (PT) or activated partial thromboplastin time (aPTT).
* Positive urine or serum pregnancy test in pre-menopausal female subjects without a documented history of surgical sterilization.
* Any concurrent serious illness that would interfere with the safety assessments including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, and hematologic disease.
* Historical Rankin score greater than or equal to 2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
rate of clot size removal | baseline to 24 hours(±12) post the last dose of rt-PA

SECONDARY OUTCOMES:
Mortality | 30 days
Procedure related mortality | 30 days
Incidence of intracranial infection | 30 days
Rate of rebleeding | 30 days
Glasgow outcome scale gos | 90 days
Glasgow outcome scale gos | 180 days
Rankin stroke impact scale | 90 days
Rankin stroke impact scale | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Suiqiang, doctor, Principal Investigator — Hubei Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Morgan T, Zuccarello M, Narayan R, Keyl P, Lane K, Hanley D. Preliminary findings of the minimally-invasive surgery plus rtPA for intracerebral hemorrhage evacuation (MISTIE) clinical trial. Acta Neurochir Suppl. 2008;105:147-51. doi: 10.1007/978-3-211-09469-3_30. PMID 19066101
- [Background] Mould WA, Carhuapoma JR, Muschelli J, Lane K, Morgan TC, McBee NA, Bistran-Hall AJ, Ullman NL, Vespa P, Martin NA, Awad I, Zuccarello M, Hanley DF; MISTIE Investigators. Minimally invasive surgery plus recombinant tissue-type plasminogen activator for intracerebral hemorrhage evacuation decreases perihematomal edema. Stroke. 2013 Mar;44(3):627-34. doi: 10.1161/STROKEAHA.111.000411. Epub 2013 Feb 7. PMID 23391763
- [Background] Lian LF, Xu F, Tang ZP, Xue Z, Liang QM, Hu Q, Zhu WH, Kang HC, Liu XY, Wang FR, Zhu SQ. Intraclot recombinant tissue-type plasminogen activator reduces perihematomal edema and mortality in patients with spontaneous intracerebral hemorrhage. J Huazhong Univ Sci Technolog Med Sci. 2014 Apr;34(2):165-171. doi: 10.1007/s11596-014-1252-x. Epub 2014 Apr 8. PMID 24710926
- [Background] Tang ZP, Shi YH, Yin XP, Xu JZ, Zhang SM, Wang W. Modifying the details of aspiration operation may contribute to the improvement of prognosis of patients with ICH. Turk Neurosurg. 2012;22(1):13-20. doi: 10.5137/1019-5149.JTN.4219-11.0. PMID 22274965